CLINICAL TRIAL: NCT00948038
Title: Dairy Modulation of Oxidative and Inflammatory Stress in Overweight and Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Dairy Management Inc. (Industry)
Responsible Party: Michael B. Zemel, Professor, The University of Tennessee
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: DMI-033
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2009-07-29 (Estimated); Status verified 2009-07

CONDITIONS: Obesity; Overweight
Keywords: Inflammation; Oxidative stress
MeSH Terms: conditions — Obesity; Overweight; Inflammation | interventions — Milk

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Soy (Active Comparator): Soy-based supplement to normal diet
  Interventions: Dietary Supplement: Soy
- Milk (Experimental): Milk-based supplement to normal diet
  Interventions: Dietary Supplement: Milk

INTERVENTIONS:
Dietary Supplement: Milk — Milk-based smoothie containing 170 kcal, 10 g protein, 1 g fat, 30 g carbohydrate adn 350 mg Ca. Three consumed each day.
  Arms: Milk
Dietary Supplement: Soy — Soy-based smoothie containing 170 kcal, 10 g protein, 1 g fat, 30 g carbohydrate and 30 mg Ca. Three consumed each day for 28 days,
  Arms: Soy

SUMMARY:
The objective of this study is to determine the acute effects of a dairy supplement compared to a soy supplement on oxidative and inflammatory stress in overweight and obese subjects in the absence of any changes in adiposity.

DETAILED DESCRIPTION:
Obesity is associated with sub-clinical chronic oxidative and inflammatory stress, both of which are major contributors to obesity-associated co-morbidities. Calcitriol (1, 25-(OH)2-D3) regulates adipocyte lipid metabolism, while dietary calcium inhibits obesity by suppression of calcitriol. We have recently shown calcitriol to increase oxidative stress and to stimulate the expression and release of inflammatory cytokines, while inhibiting the expression and release of anti-inflammatory cytokines. We have also shown that inhibition of calcitriol with high calcium diets decreases both adipose tissue and systemic oxidative and inflammatory stress in a mouse model of obesity. Moreover, dairy exerted a greater effect on both oxidative and inflammatory stress. These mice also exhibited significant reductions in adiposity, which could lead to confounding, as this reduction will independently reduce oxidative and inflammatory stress. However, the supporting cellular/mechanistic data indicate an effect which is independent of adiposity reduction. Consequently, we propose that low calcium diets exacerbate oxidative and inflammatory stress and that high dairy diets can attenuate both independently of changes in adiposity, thereby significantly reducing the risk of obesity-associated co-morbidities. Accordingly, the objective of this study is to determine the acute effects of a dairy-rich diet on oxidative and inflammatory stress in overweight and obese subjects in the absence of any changes in adiposity.

Twenty subjects (10 obese and 10 overweight) will undergo a randomized crossover study of low dairy and high dairy eucaloric diets. Each dietary period will be four weeks, and the two dietary periods will be separated by a four-week washout period. Primary outcomes will be circulating indices of oxidative stress and of inflammation. Secondary outcomes include blood pressure, circulating glucose, insulin, lipids, calcium-regulatory hormones and body composition.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 25-29.9 (n=10); 30-34.9 kg/m2 (n=10)
* Age 18-50 years
* Weight stable: no more than 3 kg weight loss during past three months

Exclusion Criteria:

* BMI < 25 or >35
* Type II diabetes requiring the use of any oral antidiabetic agent and/or insulin (because of confounding effects on ROS)
* Adverse response to study foods (lactose intolerance, dairy intolerance, dairy allergy); this will be determined by self-report.
* history or presence of significant metabolic disease which could impact on the results of the study (i.e. endocrine, hepatic, renal disease)
* history of eating disorder
* presence of active gastrointestinal disorders such as malabsorption syndromes
* pregnancy or lactation
* use of obesity pharmacotherapeutic agents within the last 6 months
* use of over-the-counter anti-obesity agents (e.g. those containing phenylpropanalamine, ephedrine and/or caffeine) within the last 6 months
* Recent (current or past 12 weeks) use of any psychotropic medication
* Recent (past four weeks) initiation of an exercise program
* Recent (past twelve weeks) initiation of hormone replacement therapy or change in HRT regimen
* Recent (past twelve weeks) initiation of hormonal birth control or change in hormonal birth control regimen
* Recent (current or past 12 weeks) history of smoking

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Plasma malondialdehyde | 28 days
Plasma 8-isoprostane F2-alpha | 28 days
Plasma tumor necrosis factor alpha | 28 days
plasma interleukin 6 | 28 days
Plasma C-reactive protein | 28 days
Plasma MCP-1 | 28-days
Plasma interleukin 15 | 28 days
Plasma adiponectin | 28 days

SECONDARY OUTCOMES:
Plasma lipids | 28 days
Plasma insulin | 28 days
vitamin D | 28 days
Body composition | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Tennessee, Knoxville, Tennessee, United States